CLINICAL TRIAL: NCT04684576
Title: Early Powered Mobility for Toddlers With Cerebral Palsy: A Comparative Case Series of the Permobil® Explorer Mini and a Modified Ride-On Car
Brief Title: Early Powered Mobility for Toddlers With Cerebral Palsy Using the Permobil® Explorer Mini and a Modified Ride-On Car
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Oregon State University (Other); Grand Valley State University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Heather Feldner, Assistant Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00011386; P2CHD101912 (NIH)
Record Dates: First submitted 2020-12-04; First posted 2020-12-24 (Actual); Results first posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy
Keywords: At risk for cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: A mixed-methods, randomized, counterbalanced 2x2 crossover intervention study. Condition A is 8-weeks of Permobil Explorer Mini Use, and Condition B is 8-weeks of modified ride-on car use.
Who Masked: Outcomes Assessor
Masking Description: The researcher who will be completing the developmental assessment scoring will be masked as to which device the child has used and when.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Explorer Mini First (AB Arm) (Experimental): Children randomized into this arm will first trial a Permobil Explorer Mini powered mobility device over an 8-week intervention period, then trial a modified ride-on car over a second 8-week intervention period in their home and community environments.
  Interventions: Device: Permobil Explorer Mini; Device: Modified Ride-On Car
- Modified Ride On Car First (BA Arm) (Active Comparator): Children randomized into this arm will first trial a modified ride-on car over an 8-week intervention period, then trial a Permobil Explorer Mini powered mobility device over a second 8-week intervention period in their home and community environments.
  Interventions: Device: Permobil Explorer Mini; Device: Modified Ride-On Car

INTERVENTIONS:
Device: Permobil Explorer Mini — The use of powered mobility devices for young children with cerebral palsy is increasingly recommended. The Permobil Explorer Mini is a new pediatric powered wheelchair that has been cleared by the FDA. The Explorer Mini will be provided for 8-weeks, and families will be provided with suggested use frequencies and provided with support for implementing the device intervention with their child.
Device: Modified Ride-On Car — Access to commercial powered mobility devices is often limited by funding or size. Many families use toy ride-on cars for early mobility, which can be easily adapted for safety and accessibility. The modified ride-on car will be provided for 8-weeks, and families will be provided with suggested use frequencies and provided with support for implementing the device intervention with their child.

SUMMARY:
The use of powered mobility devices for young children with cerebral palsy (CP) has been gaining traction, with evidence that the use of powered mobility at young ages complements (rather than detracts from) other interventions focused on more traditional mobility skills such as crawling and walking. This study will collect preliminary data (both numeric and opinion/perception data) to investigate device use patterns, caregiver perceptions, and developmental outcomes of children with CP as families are introduced to two early powered mobility interventions: the Permobil® Explorer Mini, and a modified ride-on toy car.

DETAILED DESCRIPTION:
Overview:

This study will examine how early powered mobility devices impact the lives of children with cerebral palsy (CP) and their families. Investigators will compare a modified ride-on car to one specifically designed for children 12-36 months with disabilities to understand how the early introduction of these devices affects the child's developmental outcomes, examine device use patterns (frequency, duration, and environment) and evaluate caregiver perceptions of a motorized mobility device. Research comparing these devices in natural environments will provide critical data regarding early powered mobility for children with CP.

Abstract:

Children diagnosed with CP, or children being monitored for signs and symptoms related to CP, make up the largest group of children affected by a disability. Across the lifespan, many people with CP use powered mobility devices such as scooters and wheelchairs to support their mobility and participation in home and community settings. However, the trend in early intervention has been to delay use of devices until efforts to promote independent walking are exhausted, despite strong evidence that supports early use of powered mobility to assist with participation in everyday activities. Additionally, research has indicated the use of powered mobility complements (rather than detracts from) other interventions focused on more traditional self-initiated mobility skills such as crawling and walking.

Study investigators have been involved in an international mobility and socialization program called Go Baby Go, which provides safety and accessibility modifications to commercially available toy ride-on cars. In compliment to this work, their colleagues at Permobil® have designed and recently received FDA clearance for the Explorer Mini, a powered mobility device specifically designed for children 12-36 months with disabilities such as CP to enhance their mobility and environmental exploration. Both these early powered mobility options offer functional, aesthetic, and affordable alternatives for children and families to fill a gap left by traditional powered wheelchairs.

Investigators are using a mixed-methods study to investigate the device use patterns, caregiver perceptions, and developmental outcomes of children with CP and their families. This represents the first opportunity to compare the novel device (Explorer mini) with a modified ride-on car, which has also been customized to support early self-initiated mobility in a socially inviting way. Taken together, research comparing these devices in natural environments can add critical data to the evidence base supporting early powered mobility for children with CP as a part of using multiple devices for mobility to care for those with disabilities across the lifespan. This study will also create a pilot data set from which to secure future large-scale funding to assess a wider variety of mobility devices with multiple trial sites across the country. Establishing and improving this evidence base for children with CP and their families is essential to ensure equitable access to mobility and participation experiences across the lifespan using a range of technologies to support access and facilitate achievement of key developmental skills. The aims are to: 1) Evaluate a powered mobility intervention to promote developmental, activity and participation outcomes of young children with CP; and 2) Compare the use patterns (frequency, duration, environment) of two powered mobility options: The Explorer Mini and a modified ride-on car.

ELIGIBILITY:
Inclusion Criteria:

The child will:

1. be between 12-36 months old;
2. have a medical diagnosis of CP with any level (I-V) of associated motor ability according to the Gross Motor Function Classification System (GMFCS) or be at risk for CP according to birth history and current developmental status;
3. be able to attain a seated position with or without support;
4. be able to tolerate upright sitting with or without support while moving through space for 30 minutes;
5. live in a household where English is spoken proficiently.

Adults will:

1. be 18 years or older and be the legal caregiver for the child participant;
2. demonstrate proficiency in English. Inclusion criteria will be secured via caregiver report using screening questions.

Exclusion Criteria:

Child will be excluded if:

1. they have not been given a medical diagnosis of CP or are not at risk for CP (per parent report of birth history and current developmental status);
2. if they cannot attain a seated position with or without support;
3. if they cannot tolerate upright sitting with or without support for 30 minutes;

   Adult caregivers will be excluded if:
4. they are not proficient in English (determined per screening process).

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Feldner, PT, PhD, PCS, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Grand Valley State University, Grand Rapids, Michigan
  - Oregon State University, Corvallis, Oregon
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD, including score report data from participation and developmental measures and device use reports will be made available to other researchers upon request and reported in aggregate on clinicaltrials.gov per NIH funding requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available 6 months following publication of study results.
Access Criteria: Study results and summaries will be publicly available at clinicaltrials.gov. For specific IPD, the study PI and co-investigators will review all requests for data sharing. Data will be shared for purposes of secondary analysis, contribution to a population-related database, or similar reasons that are intended to advance the evidence-based provision of family-centered care for children with disabilities.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across all three study sites between January and August 2021 via flyers posted to clinical contacts, on study recruitment websites, and on social media.
Pre-assignment Details: No enrolled participants were excluded from the study. Enrollment was balanced, 8 participants enrolled at each site. Randomization into groups (AB or BA) to determine order of device use was conducted independently at each site after enrollment.
Period: Overall Study
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 22.3 (7.2) | 20.9 (5.8) | 21.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 10 | 17
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Developmental Outcomes From Baseline to 8 Weeks
Description: The Bayley Scales of Infant Development (BSID), 4th Edition is an internationally recognized, norm referenced set of tests designed to assess developmental domains from one month to 42 months of age. This BSID-IV assessment includes Cognitive, Receptive Communication, Expressive Communication, Gross Motor, and Fine Motor subscales. Each subscale has unique score value maximums, but on all subscales, higher scores mean a better outcome. Raw score scales are in increments of 1 and range from: Cognitive (0-81); Receptive Communication (0-42); Expressive Communication (0-37); Gross Motor (0-58); Fine Motor (0-46). Mean changes in Raw Scores are reported for each domain in this summary.
Time Frame: At baseline, after first 8-week device intervention period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Number analyzed (Participants) | 12 | 12
score on a scale
  Cognitive | 5.8 (9.6) | 0.25 (11.8)
  Expressive Communication | 3.9 (2.9) | 2.8 (6.5)
  Receptive Communication | 3.9 (4.1) | 2 (4.5)
  Gross Motor | 6.3 (8.6) | 1.6 (3.1)
  Fine Motor | 4.2 (6.4) | 2.2 (5.8)

2. Primary Outcome: Change in Child Developmental Outcomes From 8 Weeks to 16 Weeks
Description: as for outcome 1
Time Frame: After second 8-week device intervention period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Number analyzed (Participants) | 12 | 12
score on a scale
  Cognitive | 1.1 (8.3) | 7.4 (11.8)
  Expressive Communication | -0.1 (2.9) | -0.5 (4.0)
  Receptive Communication | 0.4 (3.6) | 0.9 (4.4)
  Gross Motor | 1.1 (3.2) | 0.2 (6.9)
  Fine Motor | 1.8 (5.5) | 0.4 (5.7)

3. Primary Outcome: Change in Child Developmental Outcomes From Baseline to 16 Weeks
Description: as for outcome 1
Time Frame: At baseline, and after the second 8-week device period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Number analyzed (Participants) | 12 | 12
score on a scale
  Cognitive Subscale | 6.8 (7.4) | 7.7 (13.3)
  Expressive Communication Subscale | 3.8 (3.6) | 2.3 (6.2)
  Receptive Communication Subscale | 4.3 (5.3) | 2.9 (6.1)
  Gross Motor Subscale | 7.3 (7.9) | 1.8 (6.9)
  Fine Motor Subscale | 5.9 (6.2) | 2.6 (5.2)

4. Primary Outcome: Change in Child Participation and Recreational Activities From Baseline to 8 Weeks
Description: Child Engagement in Daily Life (CEDL). The CEDL is a caregiver survey tool that assesses participation in family and recreational activities and uses a 5-point Likert scale to assess frequency of participation and enjoyment of participation. The CEDL also assesses participation in self-care behaviors and uses a 5-point Likert scale to assess the degree to which the child participates in the daily self-care activities of feeding, dressing, bathing, and toileting. Scores are reported for the first section, Frequency of Participation, and the third section, Participation in Self-Care, using scaled scores validated with individuals with CP, which range between 0-100. For the remaining section (Enjoyment of Participation), only raw scores are reported, with ranges of 11-55, respectively. Higher or increased scores indicate better outcomes on all scales.
Time Frame: At baseline, after first 8-week device intervention period.
Population: In this parent reported measure, all 12 participants in each arm fully completed all items in section 1 (Frequency of Participation) and section 3 (Participation in Self Care). However, 3 participants in the AB Arm and 4 participants in the BA arm chose to leave portions of section 2 (Enjoyment of Participation) blank. Therefore, there were many items in this section that had no comparator values. Thus, we included all participants who had fully completed all items for analysis from section 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Number analyzed (Participants) | 12 | 12
score on a scale
  Frequency of Participation | 3.8 (12.1) | -0.9 (9.2)
  Enjoyment of Participation: number analyzed (Participants) | 9 | 8
  Enjoyment of Participation | -0.1 (5.3) | 2 (6.4)
  Participation in Self Care | 7.3 (10.2) | 0.3 (5.7)

5. Primary Outcome: Change in Child Participation and Self-care Activities From 8 Weeks to 16 Weeks
Description: as for outcome 4
Time Frame: After second 8-week device intervention period.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Number analyzed (Participants) | 12 | 12
score on a scale
  Frequency of Participation | 0.2 (11.0) | 2.9 (8.1)
  Enjoyment of Participation: number analyzed (Participants) | 9 | 8
  Enjoyment of Participation | 0.4 (5.3) | -1.1 (5.2)
  Participation in Self Care Activities | 2.8 (8.2) | 0.3 (6.7)

6. Primary Outcome: Change in Child Participation and Self Care Outcomes From Baseline to 16 Weeks
Description: as for outcome 4
Time Frame: At baseline, and after the second 8-week device period.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Number analyzed (Participants) | 12 | 12
score on a scale
  Frequency of Participation | 4 (4.3) | 2 (4.2)
  Enjoyment of Participation: number analyzed (Participants) | 9 | 8
  Enjoyment of Participation | 0.3 (3.6) | 0.9 (3.4)
  Participation in Self Care | 10.1 (12.6) | 0.6 (5.6)

7. Secondary Outcome: Acceptability, Intervention Appropriateness, and Feasibility of The Explorer Mini
Description: Caregivers will complete a 3-measure perceptual implementation outcome survey. All measures are 4-item, 5-point likert-scale surveys. The minimum value is 1 and the maximum value is 5 per measure. The Acceptability of Intervention Measure (AIM) is designed to measure how receptive stakeholders are to adopting an intervention, the Intervention Appropriateness Measure (IAM) is designed to measure suitability of the intervention in a given environment or circumstance, and the Feasibility of Intervention Measure (FIM) is designed to measure how possible and likely stakeholders are to adopt an intervention. Higher ratings indicate better outcomes, in this case greater acceptability, intervention appropriateness, and feasibility of adoption. Mean rankings are reported out of a 5 point scale for each section.
Time Frame: After first 8-week device intervention period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Number analyzed (Participants) | 12 | 12
score on a scale
  Acceptability of the Explorer Mini | 4.5 (0.7) | 4.3 (1.0)
  Intervention Appropriateness of the Explorer Mini | 3.8 (1.2) | 4 (1.3)
  Feasibility of Adoption of the Explorer Mini | 4.1 (0.9) | 4.1 (1.1)

8. Secondary Outcome: Acceptability, Intervention Appropriateness, and Feasibility of the Ride-On Car
Description: Caregivers will complete a 3-measure perceptual implementation outcome survey. All measures are 4-item, 5-point likert-scale surveys. The minimum score is 1 and the maximum score is 5 per measure. The Acceptability of Intervention Measure (AIM) is designed to measure how receptive stakeholders are to adopting an intervention, the Intervention Appropriateness Measure (IAM) is designed to measure suitability of the intervention in a given environment or circumstance, and the Feasibility of Intervention Measure (FIM) is designed to measure how possible and likely stakeholders are to adopt an intervention. Higher ratings indicate better outcomes, in this case greater acceptability, intervention appropriateness, and feasibility of adoption. Mean rankings are reported out of a total maximum of 5 for each section.
Time Frame: After second 8-week device intervention period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Explorer Mini First (AB Arm) | Modified Ride On Car First (BA Arm)
Number analyzed (Participants) | 12 | 12
score on a scale
  Acceptability of the Ride On Car | 3.4 (1.4) | 4.5 (0.9)
  Intervention Appropriateness of the Ride on Car | 3.0 (1.4) | 4.6 (0.7)
  Feasibility of Adoption of the Ride on Car | 3.5 (1.2) | 4.1 (1.1)

9. Other Pre Specified Outcome: Changes in Caregiver Perceptions of Powered Mobility Devices, Facilitators and Barriers to Use, and Perceptions of Their Child's Developmental Progress Between 8 Weeks and 16 Weeks.
Description: Semi-structured interviews with caregivers using an interview guide will be conducted to understand their experiences using the respective powered mobility devices, barriers encountered and solutions discovered, and perceptions of self-efficacy and behavioral capacity.
Time Frame: After second 8-week device intervention period.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in Caregiver Perceptions of Powered Mobility Devices, Facilitators and Barriers to Use, and Perceptions of Their Child's Developmental Progress Between Baseline and 8 Weeks.
Description: as for outcome 9
Time Frame: At baseline, after first 8-week device intervention period.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Child Participation and Environmental Supportiveness From 8 Weeks to 16 Weeks.
Description: Young Children's Participation & Environment Measure (YC-PEM).The YC-PEM is a caregiver survey tool that has 3 sections: home, daycare/preschool, and community, with each section assessing participation and the environment. For participation items, parents are asked how often their child has participated in different types of activities, how involved their child is when participating in activities of this type, and if parents would like their child's participation to change. For environment items, parents are asked if specific aspects of the environment facilitate or hinder their child's participation and if specific supports are available and/or adequate to support their child's participation.
Time Frame: After second 8-week device intervention period.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Device Use Frequency and Patterns
Description: Caregivers will complete a driving log that indicates the date, time, and environment of Explorer Mini (A) or modified ride-on car use (B). Caregivers will also make notes about the child's enjoyment level and general activities while using each device. To supplement caregiver reported data, automated device use data such as frequency and duration of activation, average speed, and distance traveled, will be collected either via a custom data logger (mounted on the modified ride-on car) or through integrated device systems (built-in to the Explorer Mini).
Time Frame: Through study completion at 16 weeks.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Child Participation and Environmental Supportiveness From Baseline to 8 Weeks.
Description: as for outcome 11
Time Frame: At baseline, after first 8-week device intervention period.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 8 weeks per intervention, for a total of 16 weeks
Groups:
- AB Arm (Explorer Mini First): Explorer Mini Intervention: Children randomized into this arm will first trial a Permobil Explorer Mini powered mobility device over an 8-week intervention period, then trial a modified ride-on car over a second 8-week intervention period in their home and community environments.
  Permobil Explorer Mini: The use of powered mobility devices for young children with cerebral palsy is increasingly recommended. The Permobil Explorer Mini is a new pediatric powered wheelchair that has been cleared by the FDA. The Explorer Mini will be provided for 8-weeks, and families will be provided with suggested use frequencies and provided with support for implementing the device intervention with their child.
- AB Arm (Explorer Mini First): Modified Ride On Car Intervention: Children randomized into this arm will first trial a Permobil Explorer Mini powered mobility device over an 8-week intervention period, then trial a modified ride-on car over a second 8-week intervention period in their home and community environments.
  Modified Ride-On Car: Access to commercial powered mobility devices is often limited by funding or size. Many families use toy ride-on cars for early mobility, which can be easily adapted for safety and accessibility. The modified ride-on car will be provided for 8-weeks, and families will be provided with suggested use frequencies and provided with support for implementing the device intervention with their child.
- BA Arm (Modified Ride On Car First): Modified Ride on Car Intervention: Children randomized into this arm will first trial a modified ride-on car over an 8-week intervention period, then trial a Permobil Explorer Mini powered mobility device over a second 8-week intervention period in their home and community environments.
  Modified Ride-On Car: Access to commercial powered mobility devices is often limited by funding or size. Many families use toy ride-on cars for early mobility, which can be easily adapted for safety and accessibility. The modified ride-on car will be provided for 8-weeks, and families will be provided with suggested use frequencies and provided with support for implementing the device intervention with their child.
- BA Arm (Modified Ride On Car First): Explorer Mini Intervention: Children randomized into this arm will first trial a modified ride-on car over an 8-week intervention period, then trial a Permobil Explorer Mini powered mobility device over a second 8-week intervention period in their home and community environments.
  Permobil Explorer Mini: The use of powered mobility devices for young children with cerebral palsy is increasingly recommended. The Permobil Explorer Mini is a new pediatric powered wheelchair that has been cleared by the FDA. The Explorer Mini will be provided for 8-weeks, and families will be provided with suggested use frequencies and provided with support for implementing the device intervention with their child.
Arm/Group | AB Arm (Explorer Mini First): Explorer Mini Intervention | AB Arm (Explorer Mini First): Modified Ride On Car Intervention | BA Arm (Modified Ride On Car First): Modified Ride on Car Intervention | BA Arm (Modified Ride On Car First): Explorer Mini Intervention
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04684576/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04684576/SAP_001.pdf
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04684576/ICF_002.pdf